CLINICAL TRIAL: NCT01796132
Title: Antidepressant Treatments During Pregnancy and Lactation: Prediction of Drug Exposure Through Breastfeeding and Evaluation of Drug Effect on the Neonatal Adaptation and the Development of the Young Child
Brief Title: Antidepressants During Pregnancy and Lactation: Pharmacokinetics and Clinical Implications
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University Hospital, Geneva (Other); Hospices Civils de Lyon (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Chantal Csajka, Prof PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SSRI-Milk; 320030_135650 (Other Grant/Funding Number: Swiss National Science Foundation (SNSF)); 2012-004509-29 (EudraCT Number)
Record Dates: First submitted 2013-02-04; First posted 2013-02-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Depressive Disorder; Lactation
Keywords: Depression; Lactation; Breastfeeding; Pharmacokinetics; Antidepressant
MeSH Terms: conditions — Depressive Disorder; Breast Feeding; Depression | interventions — Citalopram; Duloxetine Hydrochloride; Escitalopram; Fluoxetine; Fluvoxamine; Paroxetine; Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Pregnant and/or nursing mothers not taking a SSRI or SNRI antidepressant are recruited in a non-exposed group (Control or no SSRI/SNRI). Control group participates only in the sub-studies related to neonatal adaptation, neurodevelopment, growth and early mother-infant relationship.
- SSRI/SNRI exposure (Experimental): Pregnant and/or nursing mothers under SSRI or SNRI treatment are recruited in an exposed group (SSRI/SNRI exposure). Drug regimen including dosage, frequency and duration is not modified by the study.
  Interventions: Drug: SSRI/SNRI

INTERVENTIONS:
Drug: SSRI/SNRI — Exposed group of mothers taking one of the mentioned antidepressant drugs of the class of selective serotonin reuptake inhibitors (SSRI) or serotonin/noradrenalin reuptake inhibitors (SNRI).
  Other Names: citalopram; duloxetine; escitalopram; fluoxetine; fluvoxamine; paroxetine; sertraline; venlafaxine
  Arms: SSRI/SNRI exposure

SUMMARY:
Background: The childbearing years are a time of increased vulnerability to the onset of mood disorders in women and a high prevalence of exposure to antidepressant drugs during pregnancy and postpartum has been reported. However, the lack of information regarding the milk transfer and the safety of these drugs in breastfed infants and the related fear of adverse events for the sucking infant are some of the factors responsible for stopping prematurely breast-feeding or avoiding drug therapy. Selective serotonin reuptake inhibitors (SSRI) and selective serotonin and noradrenaline reuptake inhibitors (SNRI) are the most frequently prescribed antidepressant drugs during pregnancy and the post-partum period. They exhibit a wide interpatient variability in their concentration profiles that has been related to numerous environmental, stereochemical, demographic and genetic influences that might alter the level of exposure of breastfed newborns. Limited information is available regarding the safety of use of these antidepressant drugs during lactation, and is generally derived from small studies. A comprehensive description of their distribution and quantification in milk in a larger cohort of patients under various influences and the resulting impact on milk concentrations is lacking.

Objectives: The current proposal addresses the primary objectives of quantifying the range of concentration to citalopram, escitalopram, sertraline, fluoxetine, paroxetine, fluvoxamine, duloxetine and venlafaxine in mother plasma and breast milk in relation to genetic polymorphisms, stereochemistry, demographics and environmental factors in a large cohort of depressive mothers. This will enable to derive the exposure to the breast-fed child taking into account this variability and therefore better adjust treatment to potential influences. As secondary objectives, we will examine the neurodevelopmental outcome of a sub-set of infants subjected to SSRI/SNRI in utero and/or during breastfeeding at birth, 6, 18 and 36 months, and compared to that of a control population of infants not subjected to this treatment.

Expected Results: The proposed strategy will offer new information regarding the expected level of drug exposure associated with each or with a combination of risk factors and help for optimizing the security and rationalizing the use of antidepressant treatment in lactating women. Hence, research on the safety of use of these drugs for the developing child is an area of great public health significance.

DETAILED DESCRIPTION:
see brief summary

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to deliver in the 5 maternities involved in the study;
* Mothers under treatment by any SSRI/SNRI (fluvoxamine, fluoxetine, paroxetine, duloxetine, citalopram, escitalopram, sertraline or venlafaxine);
* Mothers who intent to breastfeed their child;
* Ability to understand and willingness to sign a written informed consent document for plasma and milk withdrawal and pharmacogenetic testing.
* For the neurodevelopment follow-up part,all babies of the Maternity of Lausanne, Morges or Geneva exposed to SSRI/SNRI will be enrolled. A control group of infants of the same socio-economic status as the subset of exposed patients will be recruited in the Maternity Hospital of Lausanne.

Exclusion Criteria:

* Mothers <18 years of age patients;
* Infants of gestational age < 34 weeks;
* Mothers giving birth to infants with major malformations;
* Inability to communicate due to language problems for the mother;
* Patients with a socio-economic context making close monitoring of the child by the mother or a relative not possible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetics of SSRI/SNRI antidepressant drugs in breast milk secretion | week 1 and week 4-6 postpartum
  The principal aim is to derive exposure to the breast-fed child by simulation while integrating influencing factors on pharmacokinetics (as genetic polymorphism, stereochemistry, demographics or environmental aspects).
  5ml blood, 10ml fore-milk and 10ml hind-milk are taken from the mother during the same feed at week 1 and week 4-6 postpartum. Antidepressant drug concentrations are determined by LC-MS/MS and milk composition by human milk analyzer.Pharmacogenetic tests are performed with PCR-Taqman on maternal blood samples and cover genes involved in the metabolism (e.g CYP) and distribution (e.g. p-Gp) of antidepressants. Simulation of antidepressant drug secretion into breast milk will take into account all this information and will be performed with non-linear mixed effects modelling techniques.

SECONDARY OUTCOMES:
Examine neonatal adaptation | delivery and week 1 postpartum
  The specific aim is to evaluate neonatal adaptation after in utero exposure to antidepressants and its relation to cord blood concentration.
  5ml blood are taken from the umbilical cord and the mother at delivery. Antidepressant drug concentrations are determined by LC-MS/MS. Finnegan Score is used to evaluate the severity of possible withdrawal or discontinuation syndrome in exposed newborns.
Examine neurodevelopment | week 1, month 6, 18 and 36 postpartum
  The specific aim is to evaluate neurodevelopment of a sub-set of infants exposed to any SSRI/SNRI in utero and/or during breastfeeding compared to a control population of infants not exposed to this treatment.
  During week 1 postpartum, somatic and neurologic state of the newborn are evaluated by a pediatrician using routine measures as well as specific tools (Dubowitz's neurologic assessment, Prechtl's general movements). At month 6,18 and 36, neurodevelopment of the infants are assessed using Hammersmith Infant Neurological Examination and Bayley Scales of Infant Development III. At the same time, mother's mental well-being is determined by using self-administered questionnaires (Edinburgh Postnatal Depression Scale, State-Trait Anxiety Inventory, Parental Sens of Competence and Revised Infant Temperament Questionnaire).
Study of growth | birth, month 6, 18 and 36 postpartum
  The specific aim is to evaluate growth of infants exposed to any of the SSRI/SNRI commercialized, compared to standardized growth charts.
  Usual infant growth information (size, body weight, head circumference) are collected routinely at birth and month 6,18,36.
Examine early mother-infant relationship | Month 6 postpartum
  The specific aim is to explore the quality of early mother-infant relationship of a sub-set of infants whose mothers are treated with SSRI/SNRI, compared to that of a control population of infants not exposed to this treatment.
  At month 6 postpartum, mother-infant relationship is evaluated by pedopsychiatrists using Care Index.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Csajka, Prof PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV)
Locations (5):
- France (2):
  - Service d'Obstétrique, Service de Néonatologie; Centre Hospitalier Universitaire Nancy, Nancy, Meurthe-et-Moselle
  - Service d'Obstétrique, Service de Néonatologie; Hospices civiles de Lyon (HCL), Lyon, Rhône
- Switzerland (3):
  - Service d'Obstétrique, Service du Développement et de la Croissance; Hopitaux Universitaires Genevois (HUG), Geneva, Canton of Geneva
  - Division de Pharmacologie Clinique, Service d'Obstétrique, Service de Néonatologie, Service de Pédopsychiatrie de liaison, Unité de Pharmacogénétique et Psychopharmacologie Clinique; Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Service d'Obstétrique, Service de Pédiatrie; Ensemble Hospitalier de la Côte (EHC), Morges, Canton of Vaud

REFERENCES:
- [Background] McNamara PJ, Abbassi M. Neonatal exposure to drugs in breast milk. Pharm Res. 2004 Apr;21(4):555-66. doi: 10.1023/b:pham.0000022401.14710.c5. PMID 15139511
- [Background] Goldman AS, Hopkinson JM, Rassin DK. Benefits and risks of breastfeeding. Adv Pediatr. 2007;54:275-304. doi: 10.1016/j.yapd.2007.03.014. PMID 17918475
- [Background] Marcus SM, Flynn HA, Blow FC, Barry KL. Depressive symptoms among pregnant women screened in obstetrics settings. J Womens Health (Larchmt). 2003 May;12(4):373-80. doi: 10.1089/154099903765448880. PMID 12804344
- [Background] Bennett HA, Einarson A, Taddio A, Koren G, Einarson TR. Prevalence of depression during pregnancy: systematic review. Obstet Gynecol. 2004 Apr;103(4):698-709. doi: 10.1097/01.AOG.0000116689.75396.5f. PMID 15051562
- [Background] Poobalan AS, Aucott LS, Ross L, Smith WC, Helms PJ, Williams JH. Effects of treating postnatal depression on mother-infant interaction and child development: systematic review. Br J Psychiatry. 2007 Nov;191:378-86. doi: 10.1192/bjp.bp.106.032789. PMID 17978316
- [Background] di Scalea TL, Wisner KL. Pharmacotherapy of postpartum depression. Expert Opin Pharmacother. 2009 Nov;10(16):2593-607. doi: 10.1517/14656560903277202. PMID 19874247
- [Background] Sie SD, Wennink JM, van Driel JJ, te Winkel AG, Boer K, Casteelen G, van Weissenbruch MM. Maternal use of SSRIs, SNRIs and NaSSAs: practical recommendations during pregnancy and lactation. Arch Dis Child Fetal Neonatal Ed. 2012 Nov;97(6):F472-6. doi: 10.1136/archdischild-2011-214239. PMID 23080479
- [Background] Horstmann S, Binder EB. Pharmacogenomics of antidepressant drugs. Pharmacol Ther. 2009 Oct;124(1):57-73. doi: 10.1016/j.pharmthera.2009.06.007. Epub 2009 Jun 27. PMID 19563827
- [Background] Baumann P, Eap CB. Enantiomeric antidepressant drugs should be considered on individual merit. Hum Psychopharmacol. 2001 Dec;16(S2):S85-S92. doi: 10.1002/hup.336. PMID 12404713
- [Background] Panchaud A, Garcia-Bournissen F, Csajka C, Kristensen JH, Taddio A, Ilett KF, Begg EJ, Ito S. Prediction of infant drug exposure through breastfeeding: population PK modeling and simulation of fluoxetine exposure. Clin Pharmacol Ther. 2011 Jun;89(6):830-6. doi: 10.1038/clpt.2011.23. Epub 2011 Apr 27. PMID 21525869
- [Background] Lobo ED, Quinlan T, O'Brien L, Knadler MP, Heathman M. Population pharmacokinetics of orally administered duloxetine in patients: implications for dosing recommendation. Clin Pharmacokinet. 2009;48(3):189-97. doi: 10.2165/00003088-200948030-00005. PMID 19385712
- [Derived] Weisskopf E, Guidi M, Fischer CJ, Bickle Graz M, Beaufils E, Nguyen KA, Morisod Harari M, Rouiller S, Rothenburger S, Gaucherand P, Kassai-Koupai B, Borradori Tolsa C, Epiney M, Tolsa JF, Vial Y, Hascoet JM, Claris O, Eap CB, Panchaud A, Csajka C. A population pharmacokinetic model for escitalopram and its major metabolite in depressive patients during the perinatal period: Prediction of infant drug exposure through breast milk. Br J Clin Pharmacol. 2020 Aug;86(8):1642-1653. doi: 10.1111/bcp.14278. Epub 2020 Apr 14. PMID 32162723